CLINICAL TRIAL: NCT05453448
Title: Higher Risk of Kidney Function Decline With Entecavir Than Tenofovir Alafenamide in Patients With HBV Related Acute-on-chronic Liver Failure: Real-World Study
Brief Title: The Renal Safety of Tenofovir Alafenamide in HBV-related Acute-on-chronic Liver Failure: Real-World Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202012708
Record Dates: First submitted 2022-06-27; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Antiviral Drugs
MeSH Terms: interventions — tenofovir alafenamide; entecavir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tenofovir alafenamide (Experimental): tenofovir alafenamide,Gilead Sciences,capsule,25 mg,once a day,Continuous use for 48 weeks.
  Interventions: Drug: tenofovir alafenamide
- entecavir (Experimental): entecavir,Fujian cosunter pharmaceutical co.LTD,capsule,0.5mg,once a day,Continuous use for 48 weeks.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: tenofovir alafenamide — Antiviral therapy
  Arms: tenofovir alafenamide
Drug: Entecavir — entecavir
  Arms: entecavir

SUMMARY:
Tenofovir alafenamide (TAF) and entecavir (ETV) are the preferred agents in patients with predisposing factors for nephrotoxicity, but few studies to date have directly compared the renal safety of the two antiviral drugs in patients with acute-on-chronic liver failure (ACLF). Hence, the investigators compared the risk of kidney function decline among patients with HBV related acute-on-chronic liver failure (HBV-ACLF) treated with ETV or TAF.From April 2020 to June 2021, a total of 272 HBV-related ACLF hospitalized patients in the Xiangya Hospital of Central South University were enrolled in this prospective study. Chronic hepatitis B was diagnosed by hepatitis B surface antigen and/or hepatitis B virus deoxyribonucleic acid (HBV-DNA) positivity for ≥6 months. ACLF was diagnosed based on the criteria proposed by the APASL Working Party. All patients received antiviral therapy with TAF (25 mg QD, n=100) or ETV (0.5mg QD, n=172), and comprehensive medical treatments. Clinical and laboratory data were collected to evaluate the progression of chronic kidney disease (CKD) .

ELIGIBILITY:
Inclusion Criteria:

* the presence of hepatitis B surface antigen (HBsAg) in the serum for at least 6 months.
* evidence of active viral replication as documented by measurable HBV DNA in the serum (≥2000IU/mL).

Exclusion Criteria:

* Less than 18 years old.
* history of ESKD or kidney transplantation.
* unknown baseline estimated glomerular filtration rate (eGFR).
* coexistence with other liver diseases such as alcoholic liver disease, autoimmune hepatitis, drug-induced liver injury, or other viral infections(hepatitis A, C, and E virus or HIV infection).
* concomitant with malignant tumor or other serious diseases affecting survival time.
* patients with missing data. follow-up period of <48 weeks.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
the survival rates without transplantation | 48 weeks
  the survival rates without transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Wenting Peng, Changsha, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng W, Gu H, Cheng D, Chen K, Wu C, Jiang C, Liu J, Peng S, Fu L. Tenofovir alafenamide versus entecavir for treating hepatitis B virus-related acute-on-chronic liver failure: real-world study. Front Microbiol. 2023 May 25;14:1185492. doi: 10.3389/fmicb.2023.1185492. eCollection 2023. PMID 37303805